CLINICAL TRIAL: NCT06985953
Title: Evaluating the Impact of TrialTalkTM; to Foster Equitable Cancer Care
Brief Title: Evaluating the Communication Between Patients and Providers in Cancer Clinics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0274; A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); UW24152 (Other: UW Madison)
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: communication
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider participants (Experimental): Cancer providers who have received TrialTalk™ training.
  Interventions: Other: TrialTalk™
- Patient participants (Experimental): Patients who are treated by a cancer provider who has received TrialTalk™ training.
  Interventions: Other: TrialTalk™

INTERVENTIONS:
Other: TrialTalk™ — TrialTalk™ is a communication tool that focuses on making the options visible and accessible while involving patients in the discussion.

SUMMARY:
This clinical trial seeks to understand patients' experiences with the healthcare team and the quality of communication between patients and doctors in cancer clinics. The main question it aims to answer is:

* Does TrialTalk™ improve communication between providers and patients?

Participants will complete questionnaires before and after their standard of care clinic visit.

DETAILED DESCRIPTION:
The online TrialTalk™ training system uses evidence-based principles and best practices for instructional design for adult learners. The system uses a four-stage learning goal framework (i.e., knowledge, skill, understanding, and application) to ensure that the training moves from rote knowledge- and skill acquisition to integration, application, ownership, and long-term memory in clinical practice. The first module introduces the TrialTalk™ framework, why it's relevant and effective to patients and providers and describes the learning goals for the rest of the course. The second module focuses on essential elements of the TrialTalk™ conversation process through examples, metaphors, and description, followed by exercises at the end of the module that solidify the basic concepts of the conversational process. The third module focuses on the essential components of the diagram, how it integrates with the conversational process, and how to use it in a patient meeting. A set of assessment and reflection questions at the end of module 3 reinforces the concepts and components of the diagram. The fourth module brings all the TrialTalk™ elements together through case studies that exemplify how the conversational process and diagram work together in different types of patient meetings (for example, a new patient versus an established patient). Assessment and reflection questions at the end of module 4 focus on integrating and using the TrialTalk™ method in practice. Learners also develop a three-day action plan to begin to use TrialTalk™ with their patients. The TrialTalk™ training system provides learning resources to physicians such as a self-assessment rubric, FAQs, a checklist, and diagram template.

TrialTalk™ intervention includes two components: provider-focused skills-based training to ensure providers' competency in using the conversational and diagrammatic aspects of TrialTalk™, and the patient-facing component, which is the TrialTalk™ tool itself, to help patients understand their prognosis and treatment options in order to make a shared informed decision about their cancer management.

ELIGIBILITY:
Inclusion Criteria - Providers:

* Hematologists, medical oncologists, or hematology/oncology fellows
* Willing to complete TrialTalk™ training

Inclusion Criteria - Patients:

* ≥ 18 years old
* have a confirmed diagnosis of cancer
* identify as Black, African American, or non-Hispanic White
* potentially eligible for a therapeutic phase I, II or III clinical trial
* can read and understand English to complete the study questionnaires
* had previous visits with the enrolled provider

Exclusion Criteria - Providers:

* providers who received previous training in the TrialTalk™ method or used it in practice before will be excluded

Exclusion Criteria - Patients:

* previous enrollment in cancer intervention clinical trial
* have moderate to severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Fidelity - Providers | Monthly for 6 months
  Fidelity to the tool by providers is measured by a 9 item qualitative questionnaire, asking how many times and how providers used TrialTalk™ when talking with their patients.
Sustainability of TrialTalk™ communication tool | 1 year
  Providers will answer a 3 item questionnaire regarding their use of TrialTalk™. Items are scored on a 5 point Likert scale, where 1 = not at all and 5 = very much. Higher scores indicate better sustainability of the tool.
Change in quality of communication | Up to 2 hours
  Patient participants will rate the quality of communication they receive from their provider. They will answer a 13 item questionnaire with a 6-point Likert scale, where 0= not done and 5 = excellent. Scores range from 0-65, with higher scores indicating better communication.
Change in trust of provider | Up to 2 hours
  Patient participants will rate how much they trust their provider using a 6 item questionnaire. Scores are on a 5-point Likert scale, where 1 = not at all and 5 = extremely. Scores range from 6-30, with higher scores indicating greater trust.
Usefulness of tool | Up to 2 hours
  Patient participants will complete a 7 item questionnaire about the visual diagram created with their provider. It is scored on a 5-point Likert scale, where 1 = not at all and 5 = extremely. Scores range from 7-35, with higher scores indicating greater usefulness.
Understanding of treatment options | Up to 2 hours
  Patient participants will answer 9 yes or no questions regarding how well they understood the options presented to them during the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Patel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Wisconsin - Madison, Madison, Wisconsin